CLINICAL TRIAL: NCT05876455
Title: Comparative Evaluation of Minimally Invasive Nonsurgical Periodontal Therapy Versus Conventional Subgingival Instrumentation in Patients With Generalized Stage 2 and 3 Periodontitis - A Randomized Controlled Trial
Brief Title: Comparative Evaluation of Minimally Invasive Nonsurgical Periodontal Therapy Versus Conventional Subgingival Instrumentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RitikaArora23
Record Dates: First submitted 2023-05-05; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Periodontitis; Subgingival Plaque
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): On the conventional non-surgical periodontal therapy side, a power-driven piezo-electric ultrasonic scaling device with scaling tips will be used the majority of the time to debride subgingival biofilm and calculus, and manual standard Gracey curette instruments (Gracey curettes Hu-Friedy, Chicago, IL, USA) will be used to remove residual deposits from the root surface.
  Interventions: Procedure: Conventional Subgingival Instrumentation
- Test Group (Active Comparator): Experimental sites designated to receive minimally invasive non-surgical periodontal therapy will undergo careful scaling and root planing under magnification (use of 3.5 X magnification loupes) with mini curettes and using an ultrasonic device with specific thin and delicate tips. These instruments will be carefully inserted through the periodontal pocket of the affected tooth to reach the root surface for debridement. Caution will be taken to preserve the stability of soft tissues.
  Interventions: Procedure: minimally invasive non-surgical periodontal therapy

INTERVENTIONS:
Procedure: Conventional Subgingival Instrumentation — On the conventional non-surgical periodontal therapy side, a power-driven piezo-electric ultrasonic scaling device with scaling tips will be used the majority of the time to debride subgingival biofilm and calculus, and manual standard Gracey curette instruments (Gracey curettes Hu-Friedy, Chicago, IL, USA) will be used to remove residual deposits from the root surface.
  Arms: Control group
Procedure: minimally invasive non-surgical periodontal therapy — minimally invasive non-surgical periodontal therapy will undergo careful scaling and root planing under magnification (use of 3.5 X magnification loupes) with mini curettes and using an ultrasonic device with specific thin and delicate tips. These instruments will be carefully inserted through the periodontal pocket of the affected tooth to reach the root surface for debridement. Caution will be taken to preserve the stability of soft tissues.
  Arms: Test Group

SUMMARY:
Background- The use of minimally invasive procedures has recently been advocated for the treatment of periodontitis, to minimize patient discomfort and maximize the healing potential. These techniques usually involve the use of magnification lenses or microscopes and small instruments which reduce the risk of tissue trauma compared with traditional instruments.

Rationale- So far only descriptive data about the clinical effects of such procedure are available and comparative studies that would include other treatment alternatives are lacking. Therefore, the aim of this study is, on split-mouth model, to compare the number of diseased sites (defined by probing depth ˃ 4 mm and bleeding on probing) after conventional subgingival instrumentation and Minimally invasive nonsurgical periodontal therapy (MINST) with the usage of special mini instruments and magnifying loupes.

Objectives- To compare sites that have residual probing depth and require further surgical intervention after undergoing the two treatment modalities.

Methods- In this split mouth randomized controlled trial, Test group will undergo non surgical therapy under magnification and using special mini bladed instruments while the control group will undergo conventional subgingival instrumentation. Reevaluation will be at 6 weeks and 3 months.

Expected outcomes- If both the groups differ in outcomes after therapy, MINST can be used to minimize the number of sites that require surgery and hence will reduce treatment costs and morbidity.

DETAILED DESCRIPTION:
Aim and objectives- The aim of this study is to evaluate the clinical outcomes after minimally invasive nonsurgical periodontal therapy versus after conventional scaling and root planing in stage 2 and stage 3 generalised periodontitis patients.

Primary Objective- 1. Comparative evaluation of number of sites with residual pocket depth > 4 mm and bleeding on pocket probing after MINST versus conventional SI at the end of 6 weeks and 3 months Secondary objective-

1. Comparative evaluation of periodontal parameters viz. probing depth, clinical attachment level, gingival recession, treatment time and patient reported outcomes after MINST versus conventional SI at the end of 6 weeks and 3 months.

Methodology- Study design- This randomized controlled trial will be conducted in the department of Periodontics, Post graduate institute of dental sciences (PGIDS), Rohtak in accordance with the ethical standards outlined in the declaration of Helsinki 1975, as revised in 2013.The study design was approved by Institutional review board, PGIDS, Rohtak and ethical acceptance applied for from the Ethical committee of PGIDS, Rohtak. Patients coming to the out patient department of Periodontics, after examination, will be included in the study if they meet the following inclusion criteria.

Randomisation- It is a split mouth study so 2 quadrants within the same arch (intra arch) in each patient will be randomly allocated to test group and control group. For the randomization process, a computer-generated list will be used to define side and treatment modality.

Participants belonging to both the groups will receive oral hygiene instructions including toothbrushing, interdental cleaning, and plaque control reinforcement at every visit.

Test group- Experimental sites designated to receive minimally invasive non-surgical periodontal therapy will undergo careful scaling and root planing under magnification (use of 3.5 X magnification loupes) with mini curettes and using an ultrasonic device with specific thin and delicate tips. These instruments will be carefully inserted through the periodontal pocket of the affected tooth to reach the root surface for debridement. Caution will be taken to preserve the stability of soft tissues.

Control group- On the conventional non-surgical periodontal therapy side, a power-driven piezo-electric ultrasonic scaling device with scaling tips will be used the majority of the time to debride subgingival biofilm and calculus, and manual standard Gracey curette instruments (Gracey curettes Hu-Friedy, Chicago, IL, USA) will be used to remove residual deposits from the root surface.

Both procedures will be performed under local anesthesia and by a single experienced periodontist. All patients will be recalled after 6 weeks and 3 months after treatment for re-evaluation and professional supra-gingival plaque control.

Primary Outcome Measures:

Number of diseased sites [ Time Frame: 6 weeks, 3 months] Difference in No of Sites with PPD (probing pocket depth) > 4 mm and BOP (bleeding upon probing)

Secondary Outcome Measures:

PPD [ [ Time Frame: 6 weeks, 3 months] Average probing pocket depth CAL [ Time Frame: 6 weeks, 3 months] Clinical attachment level REC [ Time Frame: 6 weeks, 3 months] Gingival recession Sample size-: Sample size was calculated using G power statistical software. Using probing depth reduction as the outcome to determine effect size (as determined from a previous study- Ribeiro, F.V.; Casarin, R.C.; Palma, M.A.; Junior, F.H.; Sallum, E.A.; Casati, M.Z. Clinical and patient-centered outcomes after minimally invasive non-surgical or surgical approaches for the treatment of intrabony defects: A randomized clinical trial.J. Periodontol. 2011, 82, 1256-1266), a power of 80% and error of 5%, a sample size of 18 patients was calculated. Taking into account 10% attrition rate a total of 20 patients and a total of 40 quadrants will be recruited for this split mouth study.

Data collection and statistical analysis plan- Periodontal parameters will include plaque index, periodontal probing depth (PD): the distance from the free gingival margin to the bottom of gingival sulcus, gingival recession depth (REC), clinical attachment level (CAL), bleeding on pocket probing (BOP): recorded as bleeding site 30s after probing base of sulcus. These will be assessed at six sites per tooth at baseline, 6 weeks after treatment and 3 months after treatment.

The number of sites requiring surgical intervention will be noted at the last follow up at 3 months and compared between test and control groups. The time taken for both treatment types will also be noted.

The periodontal probe (UNC-15, Hu-Friedy, Chicago, IL, USA) will be used for periodontal examination by a single periodontist. Patients' reported outcomes will be evaluated on a visual analog scale (VAS) in terms of their satisfaction and any discomfort experienced.

Statistical analysis- Data will be collected and analysed at the end of study on excel sheets. Data recorded will be processed by standard statistical analysis. All statistical analysis will be carried out using statistical software (SPSS, Version 25.0 for Windows, SPSS, Chicago, IL). The normality of distribution of data will be examined by Shapiro Wilk test. Statistical analysis will be performed according to distribution of data. Test for homogeneity of variance will also be done to select statistics. If non normal distribution, Friedman test will be applied for intra group comparison and Mann Whitney test for intergroup comparison. If data will follow normal distribution, t-tests will be used for intergroup comparison and Repeated measures ANOVA for different time points. Statistical significance level will be set at p≤0.005.

ELIGIBILITY:
Inclusion criteria-

* Systemically healthy patients having generalised Stage 2 or stage 3 periodontitis according to the American Academy of Periodontology (AAP) and the European Federation of Periodontology (EFP) periodontal classification
* A full-mouth plaque score (FMPS) and full-mouth bleeding score (FMBS) <20%, at least 5 teeth in each quadrant.

Exclusion criteria-

* pregnant or lactating
* requiring antibiotic premedication
* received antibiotic treatment in the previous 3 months
* received a course of periodontal treatment within the past 6 months
* smokers
* signs of mobility and/or traumatic occlusion

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-10 (Estimated); Primary Completion 2023-10-10 (Estimated); Study Completion 2023-11-10 (Estimated)

PRIMARY OUTCOMES:
Number of diseased sites | 6 weeks and 3 months
  Difference in No of Sites with PPD (probing pocket depth) > 4 mm and BOP (bleeding upon probing)

SECONDARY OUTCOMES:
PROBING POCKET DEPTH(PPD) | 6 WEEKS AND 3 MONTHS
  It will be measured as the distance from the gingival margin to the base of the pocket using the calibrated manual periodontal probe (PCP-UNC 15 Hu-Friedy, Chicago, IL, USA). The probe will be inserted with a firm, gentle pressure to the bottom of the pocket and maintained parallel to the vertical axis of the tooth. Measurements will be noted at 6 sites of the involved teeth- mesiobuccal, midbuccal, distobuccal, mesiolingual, distolingual and midlingual.
CLINICAL ATTACHMENT LEVEL(CAL) | 6 WEEKS AND 3 MONTHS
  It will be measured from cemento-enamel junction to base of the pocket. Measurements will be made at 6 sites of the involved tooth- mesiobuccal, midbuccal, distobuccal, mesiolingual, distolingual and midlingual. The mean clinical attachment loss over all examined surfaces will be calculated.
GINGIVAL RECESSION(REC) | 6 WEEKS AND 3 MONTHS
  Gingival recession was measured as the distance from the Cementoenamel junction(CEJ) to the gingival margin (GM), parallel to the long axis of the tooth starting from the most apical point of recession.

CONTACTS AND LOCATIONS:
Overall Officials: Ritika Arora, MDS, Principal Investigator — PGIDS,ROHTAK
Locations (1):
- Post graduate institute of dental sciences, Rohtak, Haryana, India